CLINICAL TRIAL: NCT03058926
Title: Coordinating and Data Management Center for the Consortium for the Study of Chronic Pancreatitis, Diabetes, and Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: PA16-0439; 1U01DK108328-01 (NIH)
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Chronic Pancreatitis; Diabetes; Pancreatic Cancer
Keywords: Chronic Pancreatitis; Diabetes; Pancreatic Cancer; Data Management; Protocol compliance; Regulatory compliance; Consortium studies
MeSH Terms: conditions — Pancreatitis, Chronic; Diabetes Mellitus; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine examined for biomarker evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic Pancreatitis
  Interventions: Other: Data Management and Monitoring
- Diabetes
  Interventions: Other: Data Management and Monitoring
- Pancreatic Cancer
  Interventions: Other: Data Management and Monitoring

INTERVENTIONS:
Other: Data Management and Monitoring — Clinical Research Support Center's Data Management and Multicenter Study Support (MCSS) teams responsible for monitoring protocol and regulatory compliance for all consortium studies.
  MCSS responsible for maintaining and tracking IRB approval and regulatory documents from each site throughout the life of the study.

SUMMARY:
The data management systems, auditing, and monitoring effort are supported by the MD Anderson Cancer Center Clinical Research Support Center (CRSC). The The Coordination and Data Management Center (CDMC) will provide high quality, efficient and consistent leadership and services in all aspects of data quality and assurance; data harmonization and management; while providing assistance to the projects in disseminating and interpreting those data. The CDMC PI will provide statistical (study design, analysis plans, data analysis, and interpretation), data management, and data monitoring/auditing (data quality assurance and harmonization) expertise for the proposed projects. The Cancer Center will have access to identifiable data from studies; analysis of this data will not be conducted under this protocol. Any future analysis conducted on data or specimens as part of CPDPC protocols will be conducted under a separate IRB approved data or lab protocol.

The CDMC will leverage existing support, infrastructure, and resources from the Data Management and Coordinating Center for the Global Cancer Early Detection and the clinical expertise of the Division of Pathology/Lab Medicine at MDACC.

ELIGIBILITY:
Inclusion Criteria:

* Participants with chronic pancreatis, diabetes, and pancreatic cancer recruited through Consortium.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants recruited from external sites.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2017-01-19 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Protocol and Regulatory Compliance for Consortium Studies for the Study of Chronic Pancreatitis, Diabetes, and Pancreatic Cancer (CPDPC) | 3 years
  Clinical Research Support Center's Data Management and Multicenter Study Support (MCSS) will monitor data quality and protocol compliance at all participating institutions.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org